CLINICAL TRIAL: NCT01574131
Title: Acute and Long-Term Outcome Investigations of Fenofibrate on Severely Burned Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lost funding; Shriner Burn Hosp has revoked access to study records. No updates or results can be submitted
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-106
Record Dates: First submitted 2012-03-22; First posted 2012-04-10 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2016-02

CONDITIONS: Second or Third Degree Burns
Keywords: Burn; Fenofibrate; PPAR alpha agonist; insulin sensitivity; mitochondrial
MeSH Terms: conditions — Neoplasm Metastasis; Burns; Insulin Resistance | interventions — Fenofibrate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): pill
  Interventions: Drug: Sugar Pill
- Fenofibrate (Active Comparator): ppar-alpha agonist
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — Pill 54 mg or 160 mg tablets every day for 6 months Dosing-5mg/kg up to 160 mg for 6 months
  Other Names: Lofibra
  Arms: Fenofibrate
Drug: Sugar Pill — pill every day for 6 months
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to learn the following: whether long-term treatment (6 months) with fenofibrate will decrease burn related sugar and fat increased in the blood and help prevent muscle loss and improve wound healing.

DETAILED DESCRIPTION:
Following severe burn injury in human patients the mitochondrial fat oxygenation capacity is decreased in muscle. This is associated with a corresponding progression in the severity of the resistance to the action of insulin on glucose disposal and protein synthesis and breakdown in muscle, regenerating wound and liver.

Fatty acids or their active intracellular products ( e.g. Diacylglycerol, acyl- Coenzyme A(CoA) or acylcarnitine) are the direct inhibitors of insulin action, rather than tissue triglycerides(TG) itself. In other words, impaired mitochondrial fatty acid oxygenation is the mechanism that causes altered lipid metabolism that ultimately contributes to insulin resistance.

Accumulation of active fatty acid products, such as Diacylglycerol, acyl-CoA or acylcarnitine esters in muscle cells is due to the rate of uptake of plasma free fatty acids(FFA) exceeding the rate of oxygenation within muscle due principally to a reduced capacity of mitochondria to oxidize fatty acids.

Decreasing insulin sensitivity in muscle is related to impaired insulin signaling. This will be reflected by increased activity of protein kinase C (PKC). Because PKC is thought to exert its regulatory effect primarily on either tyrosine kinase activity on the insulin receptor or downstream kinase insulin receptor substrate (IRS) phosphorylation, these elements of the insulin signaling cascade will be decreased. In turn, elements of insulin signaling related to the response of muscle glucose (PI3 Kinase) and protein (P70S6k)metabolism will be reduced. The investigators propose that increased tissue PKC activity will be associated with increased tissue concentration of Diacylglycerol, acyl-CoA or acylcarnitine. The investigators hypothesize that the treatment of patients with the peroxisome proliferator-activated receptor (PPAR) alpha antagonist fenofibrate will improve mitochondrial capacity to oxidize fatty acids. Insulin sensitivity in muscle, skin and liver in terms of both glucose and protein metabolism will be improved by fenofibrate treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥40% Burn
* ages 4-20years
* body weight ≥10kg

Exclusion Criteria:

* <40% burn
* ages <4->20 years
* body weight <10kg
* Respiratory insufficiency
* Multiple fractures
* History of cancer in last 5 years
* Bilirubin>3mg/dL
* Serum Creatinine>3mg/dL after fluid resuscitation
* Glutamyl-Oxaloacetic Transaminase(GOT) >40 Units/L
* Glutamyl-Pyruvate Transminase(GPT) >51 Units/L
* Associated head injuries requiring therapy
* Associated injuries to the chest or abdomen requiring surgery
* Receipt of any experimental drug other than the ones supplied within two months of study
* Any metal in body including rods, cardiac defibrillators, pacemaker, etc
* Orthopedic casting which would prevent placement in MRI
* Hepatitis
* Abnormal EKG
* Electrical burns

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Mitochondrial fatty acid oxygenation | 6 months post injury
  Changes in mitochondrial oxygen consumption, Palmitoyl-CoA, palmitoyl-L-Carnitine, Pyruvate, Malate, Malonyl-CoA

SECONDARY OUTCOMES:
Insulin sensitivity | 6month post injury
  Muscle amino acid uptake, protein synthesis and breakdown. Insulin receptor tyrosine kinase activity, insulin receptor substrate activity,protein kinase C activity,glucose uptake and enrichment. Fractioned synthetic rate of plasma proteins
Protein Metabolism | 6 months post injury
Glucose Metabolism | 6 months post injury
Amino Acid Metabolism | 6 months post injury

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States